CLINICAL TRIAL: NCT07277062
Title: Optimisation and Outcome Evaluation of a Just-in-time Adaptive Intervention (JITAI) for Sleep and Circadian Problems: A Micro-randomised Trial and a Randomised Controlled Trial
Brief Title: Optimisation and Evaluation of a Just-in-time Adaptive Intervention (JITAI) for Sleep and Circadian Problems (Phase I and II)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSY038
Record Dates: First submitted 2025-11-26; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Sleep and Circadian Problems
Keywords: Just-in-time Adaptive Intervention (JITAI); sleep and circadian problems; sleep-wake patterns; insomnia; sleep; ecological momentary assessment; mHealth
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The Phase II of this study uses a micro-randomized trial (MRT) design to optimise the advanced GoodShleep alongside wearable devices and EMA. Participants will participate in the JITAI through the advanced GoodShleep and will be randomly assigned to receive contextually personalised suggestions (probability 0.375), generic messages (probability 0.375), and no notifications (probability 0.3) based on our micro-randomised algorithm at a decision point.
  These notifications are intended to serve as cues to action, enhancing the participants' readiness to engage in sleep-promoting behaviours in accordance with the health belief models. The notifications will complement the 8-week, modular TranS-C intervention, which is thoroughly described in the Intervention Protocol section. All participants will receive the cross-cutting modules and core modules of TranS-C, along with selected optional modules based on the specific needs of each participant.
Masking Description: The participants and outcomes assessor will also be blinded during the micro-randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Just-in-time adaptive intervention (GoodShleep) group (Experimental): Participants will be micro-randomised to the delivery of the behavioural components at each of the 4 decision points daily, with a 37.5% chance of being micro-randomised to contextually personalised suggestions, 37.5% to generic messages, and 25% to no notifications. The randomisation process will be independent to prior randomisations and the participants' responses to previously delivered intervention suggestions.
  1. Context-based behavioural strategies based on TranS-C will be suggested through push notifications if specific decision rules are met at specific decision points.
  2. Participants will receive non-personalised standard messages instead of personalised suggestions based on the TranS-C. These messages will be sent to acknowledge their sleep problems and provide general encouragement to consider taking action to improve their conditions.
  3. This group will not receive specific notifications encouraging them to make changes.
  Interventions: Behavioral: Just-in-time adaptive intervention (JITAI) based on TranS-C (GoodShleep)

INTERVENTIONS:
Behavioral: Just-in-time adaptive intervention (JITAI) based on TranS-C (GoodShleep) — GoodShleep will comprise (1) an 8-week, smartphone-based JITAI on TranS-C; (2) EMA prompted by push notifications to detect sleep-wake regularity and mood status; and (3) 24-hour real-time wearables assessing sleep and activity.
  The TranS-C materials will be presented in text format supplemented with diagrams, video/audio clips, quizzes, and culturally relevant examples. Across the 8 sessions, 4 cross-cutting modules will be introduced, including case formulation, sleep and circadian education, motivational interviewing, and goal setting. In addition, the participants will receive 4 core modules addressing sleep-wake regularity, daytime functioning, correcting beliefs, and maintaining behavioral change. Additionally, 5 selected optional modules will be delivered based on the participant's sleep-wake features and presentations addressing sleep efficiency, excessive time in bed, delayed/advanced sleep phase, sleep-related worry, and nightmares.

SUMMARY:
The JITAI approach holds considerable promise for addressing current challenges in mHealth, including the limitations in supporting real-time monitoring, timely intervention, and poor adherence. However, research on JITAIs in the field of behavioural sleep medicine is still in its infancy. Leveraging existing pilot data, this project will entail a micro-randomised trial (MRT) designed to optimise the JITAI components and a randomised controlled trial (RCT) to examine the efficacy of the optimised JITAI on sleep and circadian functions. Specifically, research has indicated that contextually tailored suggestions are more effective in promoting health behaviors compared to generic messages. This study will include personalised, in-the-moment actionable suggestions based on the Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) to evaluate their efficacy in contrast to generic messages and no notifications.

The proposed project will have three phases. Phase I will be the technological advancement of the JITAI app, GoodShleep. Based on research findings, additional intervention engagement strategies will be added to improve adherence, including personalisation (i.e., personalised feedback and intervention content), gamification (i.e., goal setting and rewards for a completed mission), and reminders (i.e., push notifications). The refined app will be beta-tested by the research team and five individuals experiencing sleep or circadian problems to ensure the app's functionality and usability. Issues that may arise during Phase I will be resolved prior to commencing Phase II.

Phase II will be an MRT aiming to optimise the advanced GoodShleep alongside wearable devices and ecological momentary assessment (EMA). A total of 77 participants with sleep or circadian problems will participate in the JITAI through the advanced GoodShleep, which will comprise (1) an 8-week, smartphone-based JITAI on TranS-C; (2) EMA prompted by push notifications to detect sleep-wake regularity and mood status; and (3) 24-hour real-time wearables assessing sleep and activity. Participants will be randomly assigned to receive contextually personalised suggestions, generic messages, and no notifications based on our micro-randomised algorithm.

Phase III will involve an RCT to evaluate the optimised JITAI app, GoodShleep + in both short- (immediately after intervention) and medium-term (12 weeks after intervention). Eighty participants with sleep and circadian problems will be randomised into the optimised JITAI (GoodShleep+) and the care-as-usual (CAU) group in a 1:1 allocation ratio. The JITAI (GoodShleep) will be adjusted and finalised based on the findings from Phase II to transform into the optimised JITAI (GoodShleep+). The GoodShleep+ group will receive an 8-week, smartphone-based GoodShleep+ based on TranS-C. The CAU group will not receive the GoodShleep+ but will have access to usual care based on their needs and preferences. The CAU group will receive GoodShleep+ after completing all the assessments. Major assessments will be conducted at baseline, immediate post-intervention and 12-week follow-up. Participants' sleep conditions will be evaluated using the brief consensus sleep diary and wearables. Activity levels will be measured using wearables at multiple time points. Mood status will be assessed using selected items from PANAS-SF. Participants' weekly sleep and circadian functions will be monitored using Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance (SD) and Sleep-Related Impairment (SRI). Other outcomes will include sleep quality, anxiety and depression symptoms, sleep-related cognitions, overall daytime sleepiness, fatigue, quality of life and functional impairment. Intervention acceptability and intervention adherence will also be assessed.

The current registration is only for Phase I and II of the current research project.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years living in Hong Kong
* Chinese language fluency and literacy
* Experiencing ≥1 sleep or circadian problems for 3 months based on the Sleep and Circadian Problems Interview, an adapted version of the Insomnia Interview Schedule (i.e., time needed to fall asleep ≥30 minutes for ≥3 nights per week, wake after sleep onset ≥30 minutes for ≥3 nights per week, <6-hour sleep per night or ≥9-hour sleep per night per 24hour period for ≥3 nights per week, variability in the sleepweek schedule ≥2.78 hours within a week, and falling asleep after 2:00 AM on ≥3 nights per week)
* One or more PROMIS-Sleep Disturbance (PROMIS-SD) item scores ≥4 after reverse scoring
* Having adequate opportunity and circumstances for sleep to occur
* Installing the JITAI app in an Internet-enabled mobile device (iOS or Android operating system)
* Are willing to provide informed consent and comply with the trial protocol

Exclusion Criteria:

* Involving in any psychological treatment for sleep disturbances in the past 6 months
* Self-report of a significant untreated severe mental illness (e.g., bipolar disorder, psychotic disorder)
* Presence of medical or cognitive disorder(s), or side effects of medication that contribute significantly to sleep or circadian problems or make participation challenging based on the team's clinical judgement
* Working night shift (>2 nights per week) in the past 3 weeks (i.e., regularly scheduled work from 12AM to 6AM)
* Pregnancy or breastfeeding
* Having a medical or psychiatric condition where sleep restriction is deemed unsuitable due to potential worsening of the condition.

Other Criteria:

* Individuals who have sleep apnoea or periodic limb movement disorder commonly experience co-occurring insomnia will be included in the study due to the potential benefits they may derive from TranS-C
* To allow for greater generalisability, this study will not exclude those with mental disorders whose conditions are stable based on the research team's judgement
* If serious suicidal risk (i.e., Patient Health Questionnaire Item 9 score >2) is identified, the participant will be referred to the PA (a clinical psychologist) for further assessment and professional mental health services, if needed
* Medication use and changes will be recorded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System-Sleep Disturbance (PROMIS-SD) | Baseline, immediate post-intervention assessment (Week 9)
  8-item scales to assess sleep and circadian functions and impairments
Change in Patient-Reported Outcomes Measurement Information Sleep-Related Impairment (PROMIS-SRI) | Baseline, immediate post-intervention assessment (Week 9)
  8-item scales to assess sleep and circadian functions and impairments

SECONDARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) | Baseline, immediate post-intervention assessment (Week 9)
  A 19-item scale assessing sleep quality over the past month
Change in 7-day Consensus Sleep Diary | 8-week daily survey
  Records sleep time, wake time, perceived sleeping quality, and use of hypnotics on a daily basis
Change in Hospital Anxiety and Depression Scale (HADS) | Baseline, immediate post-intervention assessment (Week 9)
  A 14-item scale measuring anxiety and depression in both hospital and community settings
Change in 16-item version of the Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS-16) | Baseline, immediate post-intervention assessment (Week 9)
  A 16-item scale to assess sleep-related cognitions
Change in Epworth Sleepiness Scale (ESS) | Baseline, immediate post-intervention assessment (Week 9)
  An 8-item scale designed to evaluate overall daytime sleepiness
Change in Multidimensional Fatigue Inventory (MFI) | Baseline, immediate post-intervention assessment (Week 9)
  A 20-item instrument designed to measure fatigue symptoms
Change in Short Form (6-Dimension) Health Survey (SF-6D) | Baseline, immediate post-intervention assessment (Week 9)
  A preference-based single-index measure of the quality of life
Change in Sheehan Disability Scale (SDS) | Baseline, immediate post-intervention assessment (Week 9)
  A 5-item scale to assess functional impairment in work/school, social life and family life
Change in Treatment Acceptability/Adherence Scale (TAAS) | Baseline, immediate post-intervention assessment (Week 9)
  A 10-item scale of the willingness to utilise or recommend the intervention
Change in Credibility-Expectancy Questionnaire (CEQ) | Baseline, immediate post-intervention assessment (Week 9)
  A 6-item scale used to yield ratings of intervention credibility and the expectation of success
Change in System Usability Scale (SUS) | Immediate post-intervention assessment (Week 9)
  A 10-item scale evaluating the usability perception of an app
Change in wearable-derived rest-activity data | 8-week on a daily basis, 24 hours a day
  24-hour rest-activity data will be collected using research-grade wearables (actigraphy). Participants will be instructed to wear the device on their non- dominant wrist, 24 hours a day, for 8 consecutive weeks, with exceptions during water sports activities.

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong